CLINICAL TRIAL: NCT05622851
Title: A Randomized, Split-face Clinical Study on Comparative Ultrasound Analysis of Two Hyaluronic Acid Fillers for Midface Correction
Brief Title: Comparative Ultrasound Analysis of Two Hyaluronic Acid Dermal Fillers
Acronym: RES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLI.04.US.SL.015
Record Dates: First submitted 2022-11-07; First posted 2022-11-21 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2022-10

CONDITIONS: Volume Deficiency of the Midface

STUDY DESIGN:
Intervention Model Description: Randomized, split-face, subject-blinded, comparative
Who Masked: Participant
Masking Description: Subjects are blinded to treatment assignment to each side of their faces.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Restylane Contour (Active Comparator): Form: transparent gel of Hyaluronic Acid with the addition of lidocaine hydrochloride.
  Mode of administration: injection Dosage: at investigator's discretion for optimal outcome. Frequency and duration: injection at baseline and optional touch-up at week 4.
  Interventions: Device: Restylane Contour
- Juvederm Voluma (Active Comparator): Form: sterile, biodegradable, non-pyrogenic, viscoelastic, clear, colorless, homogenous gel implant of Hyaluronic Acid crosslinked with BDDE, formulated with lidocaine.
  Mode of administration: injection Dosage: at investigator's discretion for optimal outcome. Frequency and duration: injection at baseline and optional touch-up at week 4.
  Interventions: Device: Juvederm Voluma

INTERVENTIONS:
Device: Restylane Contour — Hyaluronic Acid dermal filler
  Arms: Restylane Contour
Device: Juvederm Voluma — Hyaluronic Acid dermal filler
  Arms: Juvederm Voluma

SUMMARY:
To assess and compare tissue aggregation and visualization of two Hyaluronic Acid fillers via ultrasound

DETAILED DESCRIPTION:
This is a randomized, split-face, subject-blinded, comparative study to assess and compare tissue aggregation and visualization of two Hyaluronic Acid fillers via ultrasound.

This study is designed to enroll and randomize approximately 15 subjects in a 1:1 ratio of treatment to Restylane Contour or Juvederm Voluma. All subjects are to have midface volume loss and contour deficiency.

Eligible subjects are randomized to receive treatment were injected by the Treating Investigator at Baseline. The method of injection is at the discretion of the Treating Investigator. A sufficient amount of product is injected to achieve optimal correction of the midface, in the opinion of the Treating Investigator and subject.

At the 4-week visit, after all study procedures for the visit are completed, treated subjects have the option of receiving a touch-up treatment to achieve optimal aesthetic improvement. At the 6-month, 9-month, and 12-month visits, similar study procedures are performed.

ELIGIBILITY:
Inclusion Criteria:

* Subject with midface volume loss and contour deficiency
* Ability of giving consent for participation in the study
* Agreement to adhere to the procedures and requirements of the study and to report to the institute on the day(s) and at the time(s) scheduled for the assessments

Exclusion Criteria:

* History of allergy or hypersensitivity to lidocaine and/or injectable hyaluronic acid
* Previous permanent or semi-permanent implant in proposed treatment area
* Previous biodegradable tissue augmentation therapy in the proposed treatment area within 12 months prior to the baseline visit
* History of other facial treatment/procedure at the study area (midface) in the previous 6 months that would potentially interfere with study injections (e.g., facial surgery, oral surgery, resurfacing, mesotherapy, lipolytic injections, botulinum toxin injections)

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Assess and compare tissue aggregation and visualization of Hyaluronic Acid fillers using ultrasound | Immediately post-treatment, 4 weeks, 6 months, 9 months, and 12 months after baseline
  Change in filler properties within the skin tissues. Filler properties include size, shape, and aggregation at different facial expressions.

SECONDARY OUTCOMES:
Evaluate subject satisfaction using self-assessment questionnaire | 4 weeks, 6 months, 9 months, and 12 months after baseline
  Percentage of response at 4 weeks, 6 months, 9 months, and 12 months, where subjects are asked about their satisfaction with treatment outcome on the midface. Scale consists of 3 preference questions (with no difference option) and 6 satisfaction questions (with strongly agree, agree, neutral, disagree, and strongly disagree).
Evaluate volume change in the treated areas using 3D imaging | 4 weeks, 6 months, 9 months, and 12 months after baseline
  Summary of total volume change in the midface measured by digital 3D photography at each visit. Total volume change corresponds to net volume change from baseline in the treated area.

CONTACTS AND LOCATIONS:
Overall Officials: Steven F Weiner, MD, Principal Investigator — The Aesthetic Clinique
Locations (1):
- The Aesthetic Clinique, Santa Rosa Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT05622851/Prot_SAP_000.pdf